CLINICAL TRIAL: NCT02732210
Title: Prospective Observational Study to Evaluate Persistence With Prolia® (Denosumab) in Postmenopausal Women With Osteoporosis in Routine Clinical Practice
Brief Title: Persistence With Prolia® (Denosumab) in Postmenopausal Women With Osteoporosis
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20101218
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Osteoporosis, Age-Related
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The objective of this study was to describe persistence with Prolia® 60 mg administered subcutaneously (SC) every 6 months (Q6M) at 12 and 24 months.

DETAILED DESCRIPTION:
The study was a multi-center, single-arm, prospective, non-interventional observational study in postmenopausal women with osteoporosis who had been treated with Prolia® for osteoporosis in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment within 4 weeks following administration of the first Prolia® (denosumab 60 mg) injection
* Received Prolia® subcutaneously for treatment of osteoporosis consistent with local (US/Canada) product label
* Subject or subject's legally acceptable representative has provided informed consent. Exclusion Criteria:
* Participation in ongoing or previous denosumab clinical trials
* Currently enrolled in another investigational device or drug study, or less than 6 months since ending another investigational device or drug study(s), or receiving other investigational agent(s)
* Contra-indicated for treatment with Prolia® according to the approved applicable local product label (US/Canada)
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenoapusal women with osteoporsis. Sampling method is Invitation to Volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 935 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2014-04-07 (Actual); Study Completion 2014-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (83):
- United States (60):
  - Research Site, Birmingham, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Hemet, California
  - Research Site, Laguna Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Murrieta, California
  - Research Site, Oxnard, California
  - Research Site, Santa Maria, California
  - Research Site, Santa Monica, California
  - Research Site, South Lake Tahoe, California
  - Research Site, Victorville, California
  - Research Site, Lakewood, Colorado
  - Research Site, Trumbull, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Sebring, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Alton, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Bettendorf, Iowa
  - Research Site, Detroit, Michigan
  - Research Site, East Lansing, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Woodbury, Minnesota
  - Research Site, Springfield, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Butler, New Jersey
  - Research Site, Dover, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Plainview, New York
  - Research Site, Asheboro, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Tabor City, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Centerville, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Middletown, Ohio
  - Research Site, Bend, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Lansdale, Pennsylvania
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Jackson, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Southlake, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Glendale, Wisconsin
  - Research Site, Madison, Wisconsin
- Canada (23):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victora, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Corunna, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Woodstock, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Jean-sur-Richelieu, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Westmount, Quebec
  - Research Site, Westmout, Quebec
  - Research Site, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Silverman SL, Siris E, Kendler DL, Belazi D, Brown JP, Gold DT, Lewiecki EM, Papaioannou A, Simonelli C, Ferreira I, Balasubramanian A, Dakin P, Ho P, Siddhanti S, Stolshek B, Recknor C. Persistence at 12 months with denosumab in postmenopausal women with osteoporosis: interim results from a prospective observational study. Osteoporos Int. 2015 Jan;26(1):361-72. doi: 10.1007/s00198-014-2871-6. Epub 2014 Sep 19. PMID 25236877
- [Background] Silverman SL, Siris E, Belazi D, Recknor C, Papaioannou A, Brown JP, Gold DT, Lewiecki EM, Quinn G, Balasubramanian A, Yue S, Stolshek B, Kendler DL. Persistence at 24 months with denosumab among postmenopausal women with osteoporosis: results of a prospective cohort study. Arch Osteoporos. 2018 Aug 7;13(1):85. doi: 10.1007/s11657-018-0491-z. PMID 30088189
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled into the study on 6 July 2011 and enrollment continued until the 935th participant enrolled on the 5 April 2012. All participants were to be observed for at least 2 years, the last subjects last reported end date was 14 April 2014.
Groups:
- Canada: Postmenopausal women with osteoporosis treated with Prolia® 60 mg administered subcutaneously every 6 months (Q6M) in routine clinical practice at study sites in Canada.
- United States: Postmenopausal women with osteoporosis treated with Prolia® 60 mg administered subcutaneously every 6 months (Q6M) in routine clinical practice at study sites in the United States.
Period: Overall Study
Arm/Group | Canada | United States
Started | 303 | 632
Completed | 218 | 338
Not Completed | 85 | 294
Not completed — Site Closed | 0 | 11
Not completed — Study Ended | 13 | 13
Not completed — Withdrawal by Subject | 28 | 87
Not completed — Lost to Follow-up | 5 | 57
Not completed — Death | 4 | 15
Not completed — Other | 35 | 103
Not completed — Missing | 0 | 8

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Canada | United States | Total
Number analyzed (Participants) | 303 | 632 | 935
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (9.2) | 71.9 (10.0) | 70.8 (9.9)
Age, Customized [Number; unit: participants]
  < 65 years | 115 | 152 | 267
  ≥ 65 to < 75 years | 102 | 216 | 318
  ≥ 75 years | 86 | 264 | 350
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 303 | 632 | 935
  Male | 0 | 0 | 0
Race [Number; unit: participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 16 | 9 | 25
  Black or African American | 0 | 9 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 285 | 601 | 886
  Other | 1 | 8 | 9
  Mixed race | 0 | 2 | 2
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 2 | 45 | 47
  Not Hispanic or Latino | 301 | 587 | 888

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Persistence With Prolia® at 12 Ponths
Description: A participant was considered persistent with Prolia® at 12 months if they received at least 2 Prolia® injections no more than 6 months plus 8 weeks (239 days) apart.
Time Frame: 12 months
Population: Full Analysis Set (all enrolled participants)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Canada | United States
Number analyzed (Participants) | 303 | 632
percentage of participants | 87.8 [83.6 to 91.3] | 81.0 [77.7 to 84.0]

2. Primary Outcome: Percentage of Participants With Persistence With Prolia® at 24 Months
Description: A participant was considered persistent with Prolia® at 24 months if they received at least 4 Prolia® injections and the length of time between any 2 consecutive Prolia® injections does not exceed 6 months plus 8 weeks (239 days).
Time Frame: 24 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Canada | United States
Number analyzed (Participants) | 303 | 632
percentage of participants | 74.9 [69.6 to 79.7] | 50.0 [46.0 to 54.0]

3. Secondary Outcome: Time to Non-persistence
Description: For non-persistent participants, time to non-persistence was calculated as the time between the date of the first injection and the date of last injection received during the period where the participant was still classified as persistent plus 6 months (183 days).
Time Frame: 24 months
Population: Full analysis set with non-persistence at 24 months
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Canada | United States
Number analyzed (Participants) | 76 | 316
months | 10.69 [6.05 to 12.86] | 12.14 [6.05 to 17.99]

4. Secondary Outcome: Number of Prolia® Injections Received
Description: The number of injections that a participant received over 24 months (including the baseline injection) regardless of when the injection was received.
Time Frame: 24 months
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: prolia injections
Arm/Group | Canada | United States
Number analyzed (Participants) | 303 | 632
prolia injections | 5.0 [4.0 to 5.0] | 4.0 [3.0 to 5.0]

5. Secondary Outcome: Percentage of Participants Satisfying Medication-taking Behavior at 12 Months
Description: Percentage of participants satisfying medication-taking behavior defined as, following the first Prolia® injection, the participant received a second Prolia® injection and the length of time between the first and the second Prolia® injection did not exceed 6 months with a grace period of ± 4 weeks.
Time Frame: 12 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Canada | United States
Number analyzed (Participants) | 303 | 632
percentage of participants | 82.2 [77.4 to 86.3] | 72.0 [68.3 to 75.5]

6. Secondary Outcome: Percentage of Participants Satisfying Medication-taking Behavior at 24 Months
Description: Percentage of participants satisfying medication-taking behavior defined as the participant received all 4 Prolia® injections and the length of time between any 2 consecutive Prolia® injections did not exceed 6 months with a grace period of ± 4 weeks.
Time Frame: 24 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Canada | United States
Number analyzed (Participants) | 303 | 632
percentage of participants | 62.7 [57.0 to 68.2] | 36.4 [32.6 to 40.3]

ADVERSE EVENTS:
Time Frame: 24 months
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Canada | United States
Serious Adverse Events (participants affected / at risk) | 27/303 | 95/632
Other Adverse Events (participants affected / at risk) | 0/303 | 0/632
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canada (N=303) | United States (N=632)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 5
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 3
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 4
Cardiac tamponade (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery embolism (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 2
Death (General disorders) | 0 | 3
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Aeromona infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 5
Clostridium difficile colitis (Infections and infestations) | 0 | 3
Device related sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 9
Pneumonia influenzal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 4
Wound infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 4
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 3
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Helicobacter test positive (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 2
Convulsion (Nervous system disorders) | 1 | 1
Dementia (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Essential tremor (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Hemiplegia (Nervous system disorders) | 1 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Neuritis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 3
Communication disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 2
Renal injury (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 2
Shoulder operation (Surgical and medical procedures) | 0 | 1
Spinal operation (Surgical and medical procedures) | 0 | 1
Toe amputation (Surgical and medical procedures) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 3
Hypertensive emergency (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 2
Venous thrombosis limb (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.